CLINICAL TRIAL: NCT02409056
Title: Putting CDSMP to Work: Implementation of the Live Healthy, Work Healthy Program
Brief Title: Putting CDSMP to Work
Acronym: WorkCDSMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: YMCA (Other)
Responsible Party: Principal Investigator, Mark Wilson, Associate Dean for Academic Affairs, University of Georgia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: UGeorgia
Record Dates: First submitted 2015-03-03; First posted 2015-04-06 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Chronic Disease; Cardiovascular Diseases
Keywords: intervention; translation; workplace; CVD; CDSMP
MeSH Terms: conditions — Chronic Disease; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- workplace-tailored CDSMP (Experimental): Group will receive the CDSMP program which has been modified to fit the unique characteristics of the workplace.
  Interventions: Behavioral: Workplace-tailored CDSMP
- CDSMP usual care (Active Comparator): Group will receive the standard CDSMP program which is currently being offered in a variety of community settings.
  Interventions: Behavioral: Chronic Disease Self-Management Program
- control (No Intervention): Group will receive no intervention for the first 6 months (pre / post), then be randomly assigned to one of the above interventions.

INTERVENTIONS:
Behavioral: Workplace-tailored CDSMP — This is the CDSMP program which has been modified to fit the unique characteristics of the workplace and will be offered in worksites.
  Other Names: Live Healthy Work Healthy Program
  Arms: workplace-tailored CDSMP
Behavioral: Chronic Disease Self-Management Program — This is the standard CDSMP which has been implemented in community settings.
  Other Names: CDSMP
  Arms: CDSMP usual care

SUMMARY:
This project is the test of the effectiveness of the Chronic Disease Self-Management Program which will be translated to a worksite setting.

DETAILED DESCRIPTION:
This project will test adaptations of the Chronic Disease Self-Management Program (CDSMP) designed to increase the likelihood of widespread use in workplace settings. CDSMP, which has been proven efficacious in community trials, is a six-week program that is designed to help individuals better manage their chronic disease and its many complications. Although there is considerable interest among worksite health promotion practitioners for a chronic disease program, CDSMP has not been adapted and tested in workplace settings. In this study, we will determine a) if the CDSMP program tailored to worksites can be efficacious, b) the comparative effectiveness of the worksite tailored CDSMP when compared to the original CDSMP and c) the cost-effectiveness (average and incremental) and return on investment of the two interventions. The participating sites are seven organizations from a rural county in Southwest Georgia. Our partner for the project is the local YMCA. YMCA staff will be trained to implement the program which will foster sustainability. Participants will be randomly assigned to 1) workplace-tailored CDSMP, 2) 'usual care' CDSMP, and 3) control group. Data will collected at baseline, 6-month follow-up and 12-months follow-up. The control group will be a delayed intervention group that will be randomly assigned to an intervention group after taking the 6 month survey. The primary outcome measures include blood pressure, cholesterol, blood glucose, BMI, diet, physical activity and tobacco use and the secondary measures including patient-provider communication, quality of life, medical adherence, and work performance and productivity. An average cost-effectiveness analysis will compare interventions to control and an incremental cost-effectiveness analysis will be conducted comparing each intervention to one another. The hypotheses will be tested using a growth modeling approach examining changes over time. This will enable us to maximize the dissemination and implementation of CDSMP across worksite populations by using approaches which are realistic for most work organizations.

ELIGIBILITY:
Inclusion Criteria:

* The primary target is all employees 45 years or above with levels of gender and ethnicity similar to those found in the workplaces with which we will work.
* If younger individuals wish to participate, we will not turn them away but the program is designed for older adults. It is unlikely we will get a substantial number of participants over 45.

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Body Mass Index examining change at 6 and 12 months | baseline, six months, one year
  Measure of obesity using height and weight
blood pressure examining change at 6 and 12 months | baseline, six months, one year
  diastolic and systolic measures
Cholesterol levels examining change at 6 and 12 months | baseline, six months, one year
  HDL, LDL, and total cholesterol levels
blood glucose examining change at 6 and 12 months | baseline, six months, one year
  blood glucose levels
Cardiovascular risk scale examining change at 6 and 12 months | baseline, six months, one year
  Overall measure taken from the Framing Heart Study which includes: systolic blood pressure, total cholesterol, HDL cholesterol, BMI, gender, age, use of antihypertensive treatment, smoking and diabetes mellitus status.
Eating behaviors (Food propensity questionnaire) examining change at 6 and 12 months | baseline, six months, one year
  Food propensity questionnaire used to estimate usual intake for food items and food groups.
Physical activity (Measure of moderate-intensity physical activities) examining change at 6 and 12 months | baseline, six months, one year
  Measure of moderate-intensity physical activities.
Sedentary behavior (Measures total time spent sitting in transport, work and leisure) examining change at 6 and 12 months | baseline, six months, one year
  Measures total time spent sitting in transport, work and leisure.
Tobacco use examining change at 6 and 12 months | baseline, six months, one year
  Measure of current and past tobacco use.

SECONDARY OUTCOMES:
Patient-provider communication (Measure of communication with a physician) examining change at 6 and 12 months | baseline, six months, one year
  Measure of communication with a physician.
Self-assessed quality of life scale examining change at 6 and 12 months | baseline, six months, one year
  CDC Healthy Days quality of life measure.
Depression (Personal Health Questionnaire Depression Scale (PHQ8) examining change at 6 and 12 months | baseline, six months, one year
  Personal Health Questionnaire Depression Scale (PHQ8).
Prescription medication adherence examining change at 6 and 12 months | baseline, six months, one year
  Measures medication compliance.
Pain (Visual analogue scale) examining change at 6 and 12 months | baseline, six months, one year
  Visual analogue scale to determine symptoms of chronic disease.
Sleep (Visual analogue scale) examining change at 6 and 12 months | baseline, six months, one year
  Visual analogue scale to determine symptoms of chronic disease.
Stress (Visual analogue scale) examining change at 6 and 12 months | baseline, six months, one year
  Visual analogue scale to determine symptoms of chronic disease.
Fatigue (Visual analogue scale) examining change at 6 and 12 months | baseline, six months, one year
  Visual analogue scale to determine symptoms of chronic disease.
Well-being (SF-12) scale examining change at 6 and 12 months | baseline, six months, one year
  Measure of functional health and well-being (SF-12).
Quality of life (EQ-5D) scale examining change at 6 and 12 months | baseline, six months, one year
  Measure of quality of life (EQ-5D).

OTHER OUTCOMES:
Absenteeism scale examining change at 6 and 12 months | baseline, six months, one year
  Measures absence, lateness, and performance.
Presenteeism (Work Limitations Questionnaire (WLQ) examining change at 6 and 12 months | baseline, six months, one year
  Work Limitations Questionnaire (WLQ) assess the degree to which health problems interfered with job activities.
Work ability index examining change at 6 and 12 months | baseline, six months, one year
  Assess physical and mental demands of work and worker's health status and resources.
Job satisfaction question examining change at 6 and 12 months | baseline, six months, one year
  Measures job satisfaction.
Organizational commitment scale examining change at 6 and 12 months | baseline, six months, one year
  Measures organizational commitment.
Turnover intention question examining change at 6 and 12 months | baseline, six months, one year
  Measures likelihood of leaving the organization.
Job stress scale examining change at 6 and 12 months | baseline, six months, one year
  Measures job-related stress.
Fatigue (Work-related fatigue assessment scale.) examining change at 6 and 12 months | baseline, six months, one year
  Work-related fatigue assessment scale.
Healthcare utilization (Self-report measures) examining change at 6 and 12 months | baseline, six months, one year
  Self-report measures of physician and hospital services.

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Wilson, HSD, Principal Investigator — University of Georgia; Matthew L Smith, PhD, Principal Investigator — Texas A&M University
Locations (13):
- United States (13):
  - Madison County Schools, Danielsville, Georgia
  - City of Moultrie, Moultrie, Georgia
  - Colquitt County Government, Moultrie, Georgia
  - Colquitt County Schools, Moultrie, Georgia
  - Colquitt Regional Medical Center, Moultrie, Georgia
  - National Beef, Moultrie, Georgia
  - Southwest Georgia Bank, Moultrie, Georgia
  - Southwest Georgia Community Action Council, Moultrie, Georgia
  - Southwest Regional Technical College, Moultrie, Georgia
  - Turning Point Hospital, Moultrie, Georgia
  - Lowndes County, Valdosta, Georgia
  - Valdosta City Schools, Valdosta, Georgia
  - Wiregrass Technical College, Valdosta, Georgia